CLINICAL TRIAL: NCT03472105
Title: Short-term Effect of a New Nordic Renal Diet on Phosphorus Homeostasis in CKD Stage 3-4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H-16033940
Record Dates: First submitted 2018-03-13; First posted 2018-03-21 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Chronic Kidney Disease, Stage 3 (Moderate)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: The aim of this study was to investigate if 7 days of dietary intake of New Nordic Renal Diet reduces the 24-hour urinary phosphorus excretion and other components of the phosphorus homeostasis in 18 moderate CKD patients compared to 7 days of habitual diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habitual diet (Other): 18 participants were on a habitual diet for 7 days
  Interventions: Dietary Supplement: New Nordic Renal Diet
- New Nordic Renal Diet (Active Comparator): 18 participants were given a New Nordic Renal Diet for 7 days
  Interventions: Dietary Supplement: New Nordic Renal Diet

INTERVENTIONS:
Dietary Supplement: New Nordic Renal Diet — One week ingesting a phosphorus reduced diet containing a total of 850 mg of phosphorus/day compared to one week of a habitual diet
  Other Names: Habitual Diet

SUMMARY:
Hyperphosphatemia is a severe complication to chronic kidney disease (CKD) and is associated with increased risk of vascular calcification, cardiovascular morbidity and mortality. Early dietary intervention and improvement in dietary therapy might optimally reduce cardiovascular complications. For this purpose the investigators investigated patients with CKD stage 3-4, the participants dietary habits, developed a New Nordic Renal Diet and investigated the short term effect on phosphorus homeostasis.

DETAILED DESCRIPTION:
Development of the New Nordic Renal Diet The NND was not suitable for CKD patients in its present form because of too high phosphorus content. By going through the diet composition in details and reducing some of the phosphorus rich food items such as nuts, dairy products, rye bread and fish and reducing the daily intake of meat to a total of 120 mg/day we designed the NNRD with a total of 850 mg phosphorus per day and 0.8 g protein per kg per day. Two main principles were important; affordable and palatable.

Phosphorus content of the meals The nutrient content of the meals were based on information from the Danish food composition data bank; Dankost 3000® (version 7.01, 2009, Dankost, Copenhagen, Denmark). The diets during the intervention were designed to be iso-caloric. The phosphorus content in the samples was determined by inductively coupled plasma mass spectrometry (ICPMS) at the National Food Institute at the Technical University of Denmark. Briefly, the samples were lyophilized and homogenized to a fine powder. Subsamples (0.3 g) were digested with concentrated nitric acid in a microwave oven (Multiwave 3000, Anton Paar, Graz, Austria). The quantification of phosphorus (31P) was done with external calibration using 45Sc as internal standard. The ICPMS (Thermo iCAPq, Bremen, Germany) was run in KED mode using helium as cell gas. For quality assurance of the results, the certified reference material BCR63R (Skim milk powder) was analyzed and the obtained results (10.9+/-0.3 mg/g) were in good agreement with the certified target value (11.1+/-0.13 mg/g).

Study Nineteen patients were recruited from the outpatient clinic at the Department of Nephrology, Copenhagen University, Rigshospitalet and 1 patient from Department of Nephrology, Copenhagen University, Herlev Hospital.

This was a randomized controlled crossover study of two diets in patients with CKD stage 3-4 (figure 1). Baseline data (day 0) was obtained including 24-h urine collection, fasting blood samples and dietary record. During the intervention the participants received our phosphorus reduced version of the NND termed the NNRD for 1 week, fasting blood samples was achieved on day 1 and 4 together with 24-hour urine collection. During the control period the participants kept to their habitual diet from day 1 - 6 (on day 1 and day 4, they kept a dietary record and collected 24-h urine) and on day 7 they received a control diet with a phosphorus content in accordance with an average Danish diet (1500 mg). On day 7, in both the two intervention periods, the patients were admitted to the Department of Nephrology, University Hospital of Copenhagen, Rigshospitalet to follow the circadian rhythm of plasma phosphate, plasma intact FGF23, plasma calcium and plasma PTH. Fasting blood sample and 24-h urine collection was obtained, and blood was additionally drawn 30 min after each of the three meals.

During the NNRD intervention there were two daily meals, given with a two-day rotation. Diet planning and analysis was initially done using the Food Composition Data bank (version 7.01, 2009, Copenhagen, Denmark). The actual measured phosphorus content was equal to the calculated value from the Food Composition Data bank and the diets were kept unchanged.

Self-reporting questionnaire The dietary compliance, satisfaction and satiation were judged by written self-reported questionnaire during the NNRD (supplemental material). Dietary satisfaction was judged by a five-level Likert scale with following response options: very good, good, okay, not good and bad. A similar method was used for the dietary compliance with the following response options: 100%, 80%, 60%, 40% and 20%. The satiation was judged by yes or no.

ELIGIBILITY:
Inclusion Criteria:

* Estimated glomerular filtration rate (eGFR) 16 to 45 ml/min/1.73 m2, as judged by CKD-EPI equation
* Medically stable for 2 months before and during the study
* No food allergies
* Ability to understand the Danish language orally and in writing

Exclusion Criteria:

- Intake of phosphate binders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
24-hour urine phosphorus excretion | 7 days
  primary outcome was measured by 24-hour urine collection

CONTACTS AND LOCATIONS:
Locations (1):
- Arne V. Astrup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No